CLINICAL TRIAL: NCT04113343
Title: A Phase 1 Study to Determine the Single-dose Pharmacodynamics, Pharmacokinetics, and Safety and Tolerability of Remimazolam Following Oral Administration With and Without Alcohol in Healthy Female Subjects
Brief Title: Oral Remimazolam With and Without Alcohol in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CNS7056-020
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Safety Issues
Keywords: remimazolam
MeSH Terms: interventions — remimazolam; Ethanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment A: remimazolam (Active Comparator): Oral administration of 360 mg remimazolam
  Interventions: Drug: Remimazolam
- Treatment B: remimazolam + 5% v/v alcohol (Experimental): Oral administration of 360 mg remimazolam and 5% v/v alcohol
  Interventions: Drug: Remimazolam; Other: Alcohol
- Treatment C: remimazolam + 15% v/v alcohol (Experimental): Oral administration of 360 mg remimazolam + 15% v/v alcohol
  Interventions: Drug: Remimazolam; Other: Alcohol
- Treatment D: remimazolam + 40% v/v alcohol (Experimental): Oral administration of 360 mg remimazolam + 40% v/v alcohol
  Interventions: Drug: Remimazolam; Other: Alcohol
- Treatment E: placebo + 40% v/v alcohol (Placebo Comparator): Oral administration of Placebo + 40% v/v alcohol
  Interventions: Other: Alcohol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam via oral administration
  Other Names: CNS7056
  Arms: Treatment A: remimazolam; Treatment B: remimazolam + 5% v/v alcohol; Treatment C: remimazolam + 15% v/v alcohol; Treatment D: remimazolam + 40% v/v alcohol
Other: Alcohol — Alcohol
  Arms: Treatment B: remimazolam + 5% v/v alcohol; Treatment C: remimazolam + 15% v/v alcohol; Treatment D: remimazolam + 40% v/v alcohol; Treatment E: placebo + 40% v/v alcohol

SUMMARY:
A Phase 1 Study to Determine the Single-dose Pharmacodynamics, Pharmacokinetics, and Safety and Tolerability of Remimazolam Following Oral Administration With and Without Alcohol in Healthy Female Subjects

DETAILED DESCRIPTION:
Evaluating the potential for additive or synergistic effects of alcohol when coadministered with remimazolam. Female subjects were selected because they represent the population at greatest risk for victimization in drug-facilitated sexual assault. In addition, females have a slower ethanol metabolism, therefore, the effects of remimazolam, if coadministered with alcohol, may last longer. Hence, this population represents the worst-case scenario in evaluating the risk of remimazolam misuse in drug-facilitated assault.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the trial, give written informed consent prior to the initiation of any protocol-specific procedures, and comply with the trial restrictions.
2. Able to speak, read, and understand English sufficiently to allow completion of all Trial assessments.
3. Gender : female
4. Age : 21 to 45 years, inclusive
5. Weight : ≥ 50 kg
6. Body mass index (BMI) : 18.0 to 33.0 kg/m2, inclusive
7. Healthy status, defined by the absence of evidence of any clinically significant, in the opinion of the Investigator, active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiograms (ECG), hematology, blood chemistry, serology, and urinalysis.
8. Current alcohol user classified as a moderate drinker, defined as drinking > 2 drinks/week and ≤ 14 drinks/week (1 drink equals approximately 12 oz/350 mL of beer, 5 oz/150 mL of wine, or 1.5 oz/45 mL of spirits).6
9. Ability and willingness to abstain from alcohol, caffeine, and xanthine-containing beverages or food (eg, coffee, tea, cola, chocolate, energy drinks) from 48 hours (2 days) prior to admission to the clinical facility on Day -1 until trial discharge.
10. All values for hematology and for clinical chemistry tests of blood and urine within the normal range or showing no clinically relevant deviations, as judged by the Investigator.
11. A negative pregnancy test at Screening and Day -1.
12. Females of childbearing potential must have agreed to use 2 forms of contraception, one of which must have been a barrier method, during the trial and for 90 days after the last drug administration. Acceptable barrier forms of contraception were condom and diaphragm. Acceptable nonbarrier forms of contraception for this trial were oral contraceptives, injectable hormone contraceptives, implantable birth control, intrauterine devices, and/or spermicide. Injectable hormonal contraception was allowable as a nonbarrier method.
13. Females who were not of childbearing potential, including postmenopausal females (defined as 12 months with no menses prior to Screening and a serum follicle-stimulating hormone [FSH] > 40 IU/L at Screening) or females who were surgically sterilized.

Exclusion Criteria:

1. Females who were pregnant or lactating.
2. Known intolerance towards alcohol (symptoms could include nausea, flushed face, vomiting, or hypotension upon drinking) or known alcohol dehydrogenase deficiency.
3. of Asian descent (one or both parents) due to potential for genetic polymorphism related to aldehyde dehydrogenase deficiency.
4. History of alcohol abuse or drug addiction (except nicotine or caffeine), as defined by the Diagnostic and Statistical Manual of Mental Disorders, fifth edition, text Revision (DSM-V-TR), or any self-reported dependence or "addiction" within the subject's lifetime (except nicotine or caffeine).
5. History of relevant food allergies.
6. Use of any investigational drug or device within 30 days of the first dose of Trial medication.
7. Any disease which, in the opinion of the Investigator, posed an unacceptable risk to the subjects.
8. Known allergy, hypersensitivity, or prior intolerance to benzodiazepine derivatives or flumazenil, or a medical condition such that these agents were contraindicated.
9. Use of tobacco products within 60 days prior to the first drug administration.
10. Routine or chronic use of more than 3 grams of acetaminophen daily.
11. History of donation or loss of more than 450 mL of blood or blood products within 60 days prior to dosing in the clinical research center or planned donation before 30 days had elapsed since intake of trial drug in the current trial.
12. Positive screening test for hepatitis B surface antigen (HBsAg), anti-hepatitis C Virus (HCV) antibodies, or anti-human immunodeficiency virus (HIV) 1 and 2 antibodies.
13. Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) at Screening and admission to the clinical research center.
14. Average intake of > 14 drinks of alcohol per week (1 drink equals approximately 12 oz/350 mL of beer, 5 oz/150 mL of wine, or 1.5 oz/45 mL of spirits).
15. Required concomitant treatment with any prescription or non-prescription medications (with the exception of hormonal contraceptives, hormone replacement, and acetaminophen) or natural health products (herbal remedies), or respiratory depressants, or could not safely discontinue these medications at least 7 days prior to receiving trial drug.
16. Inability to be venipunctured or to tolerate venous access, as determined by the Investigator or designee.
17. History of clinically significant, recent/current, and nonremote suicidal ideations or suicide attempts that, in the opinion of the Investigator, posed an unacceptable risk to the subject for participating in the trial.
18. Any major surgery within 4 weeks of trial drug administration. NOTE: Any parameter/test could be repeated at the Investigator's discretion during Screening and/or on Day -1.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Paired Associates Learning (PAL) Test | Predose to 4 hours postdose
  PAL Test was conducted using the software CANTAB (Cambridge Cognition)
Modified Observer Assessment of Alertness/Sedation (MOAA/S) | Predose to 4 hours postdose
  The MOAA/S scale is a validated, 6-point rating scale that involves an observer rating subjects' responsiveness to stimuli of increasing intensity (5 = alert, 0 = sedated).
Alertness/Drowsiness Visual Analog Scale (VAS) | Predose to 4 hours postdose
  The Alertness/Drowsiness VAS was administered as a 100-point bipolar scale, with 50 being the neutral point, as follows:0: Very drowsy, 50: Neither drowsy nor alert, 100: Very alert
Reaction Time Test (RTI) | Predose to 4 hours postdose
  RTI was conducted using the software CANTAB (Cambridge Cognition).
Maximum observed plasma concentration (Cmax) | Predose to 8 hours postdose
Time to Maximum observed plasma concentration (Tmax) | Predose to 8 hours postdose
Area under the plasma concentration-time curve (AUC) from zero to the last measurable concentration | Predose to 8 hours postdose
Terminal elimination half-life (T1/2) | Predose to 8 hours postdose
Apparent oral clearance (CL/F) | Predose to 8 hours postdose
Apparent volume of distribution at terminal Phase (Vz/F) | Predose to 8 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Ahad Sabet, MD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA Health Sciences (PRA) - Early Development Services, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pesic M, Stohr T, Ossig J, Borkett K, Donsbach M, Dao VA, Webster L, Schippers F. Remimazolam Has Low Oral Bioavailability and No Potential for Misuse in Drug-Facilitated Sexual Assaults, with or Without Alcohol: Results from Two Randomised Clinical Trials. Drugs R D. 2020 Sep;20(3):267-277. doi: 10.1007/s40268-020-00317-0. PMID 32757149